CLINICAL TRIAL: NCT06107647
Title: Prospective Comparisons of Active Air Blow Heaters and Resistive Type Heaters in High-current and Low-current Inhalation Anesthesia in Terms of the Prevention of Hypothermia
Brief Title: Comparisons of Two Different Type Heater in Different Inhalation Anesthesia in Terms of Prevention of Hypothermia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Abdullah Pabucci, Assistant Doctor, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ABDULLAHPABUCCI1
Record Dates: First submitted 2023-08-17; First posted 2023-10-30 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Anesthesia; Hypothermia; Heat
Keywords: High flow; hypothermia; low flow; rhinoplasty
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- GRUP DA (Experimental): Patients who will be given low-flow anesthesia during the operation and will be heated with an active air blower heater.
  Interventions: Device: COVIDIEN WarmTouch
- GRUP YA (Experimental): Patients who will be given high current anesthesia during the operation and will be heated with an active air blower heater.
  Interventions: Device: COVIDIEN WarmTouch
- GRUP DR (Experimental): Patients who will be given low-flow anesthesia during the operation and will be heated with a resistive heater
  Interventions: Device: COVIDIEN WarmTouch
- GRUP YR (Experimental): Patients who will be treated with high-flow anesthesia and heated with a resistive heater during the operation
  Interventions: Device: COVIDIEN WarmTouch

INTERVENTIONS:
Device: COVIDIEN WarmTouch — "COVIDIEN WarmTouch will be used as an active air blowing heater. Patients will be warmed starting from the beginning of anesthesia."
  "The INDITHERM Medical Alpha, which is a resistive heater, will be applied to patients starting at the beginning of anesthesia."
  Other Names: INDITHERM Medical Alpha

SUMMARY:
Unintentional perioperative hypothermia is a common occurrence. One of the recommendations of the guidelines to prevent hypothermia is the use of active warmers. It is known that low-flow anesthesia protects from hypothermia compared to high-flow anesthesia. In this study, we aimed to compare the efficacy of using active air blown heater and resistive heater in preventing hypothermia in patients with low flow and high flow inhalation anesthesia

DETAILED DESCRIPTION:
ABSTRACT

PROSPECTIVE COMPARISON OF ACTIVE AIR BLOWN HEATER AND RESISTIVE TYPE HEATERS FOR PREVENTION OF HYPOTHERMIA IN HIGH CURRENT AND LOW CURRENT INHALATION ANESTHESIA

Aim: Unintentional perioperative hypothermia is a common occurrence. One of the recommendations of the guidelines to prevent hypothermia is the use of active warmers. It is known that low-flow anesthesia protects from hypothermia compared to high-flow anesthesia. In this study, we aimed to compare the efficacy of using active air blown heater and resistive heater in preventing hypothermia in patients with low flow and high flow inhalation anesthesia.

Materials and Methods: After ethics committee approval (Date: 08.12.2022/23), 112 patients with American Society of Anesthesiologist (ASA; American Society of Anesthesiologists) I-III, who were to undergo rhinoplasty between June 01, 2023 and January 01, 2024, were included in the study after informed consent was obtained. Group DA was defined as low flow anesthesia and active air blast heater, group DR as low flow anesthesia and resistive heater, group YA as high flow anesthesia and active air blast heater, and group YR as high flow anesthesia and resistive heater. Each group consisted of 28 patients. Heart rate, systolic, diastolic and mean arterial pressure, peripheral oxygen saturation values and body temperature values were measured and recorded at certain time intervals during the perioperative period and in the recovery unit. Body temperatures were also recorded in the ward. Thermal comfort scores were evaluated on admission, in the recovery unit and in the ward, while shivering score and patient satisfaction score were evaluated only in the recovery unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-65, who are included in the ASA I-III group, who will undergo rhinoplasty.

Exclusion Criteria:

* Patients with BMI > 35 KG/M²
* Patients with body temperature >37.5°C, <36°C degrees
* Those with cardiovascular system or central nervous system disease
* Patients with thyroid disorders
* Patients with autonomic dysfunction
* Patients not between the ages of 18-65
* Patients with missing information in the information form
* Patients using steroids or vasoactive drugs.
* Patients whose operation time is less than 30 minutes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of body temperatures in patients using two different body heaters during anesthesia applications. | 6 mounth
  In our study, two patient groups receiving high current and low current anesthesia will be heated with only one type of heater, either active air blowing heater or resistive heater, from the beginning of anesthesia. Their body temperatures will be measured and recorded throughout the operation.
  In our study, COVIDIEN WarmTouch will be used as an active air blowing heater. INDITHERM Medical Alpha will be used as a resistive-type heater. Throughout the entire operation, body temperature will be monitored using the zero-heat flow method from the temporal artery to the body surface (3M Spot ON).

CONTACTS AND LOCATIONS:
Overall Officials: abdullah pabucci, Principal Investigator — fatih sultan mehmet research and traning hospital
Locations (1):
- Abdullah Pabucci, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No